CLINICAL TRIAL: NCT06579391
Title: Effects of a Targeted Nutritional Supplement on Muscle Volume and Function After Posterior Lumbar Spine Surgery: A Randomized, Placebo-Controlled, Double-Blind Clinical Trial
Brief Title: Targeted Nutritional Supplement After Lumbar Spine Surgery: A Randomized, Placebo-Controlled, Double-Blind Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Institutional barriers.
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Sohaib Zafar Hashmi, Assistant Clinical Professor, Department of Orthopaedic Surgery, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2811
Record Dates: First submitted 2024-03-31; First posted 2024-08-30 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Lumbar Spinal Stenosis
Keywords: nutritional supplementation; essential amino acids; lumbar spine surgery; paraspinal muscle volume; paraspinal muscle fatty infiltration
MeSH Terms: conditions — Spinal Stenosis | interventions — Amino Acids, Essential; Alanine

STUDY DESIGN:
Intervention Model Description: This is a two-arm, randomized, placebo-controlled, double-blinded, single-center clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): One scoop (20 grams) of EAAs mixed in 10-12 ounces of a cold beverage to taste preference consumed orally twice daily between meals for 1 week before surgery up until 2 weeks after surgery.
  Active ingredients: L-leucine (3.6g), L-lysine as L-lysine HCl (3.2g), L-phenylalanine (3.2g), L-valine (2.4g), L-threonine (2.8g), L-isoleucine (2.0g), L-methionine (0.6g), and L-histidine as L-histidine HCl (2.2g)
  Interventions: Dietary Supplement: Essential amino acids
- Placebo (Placebo Comparator): One scoop (20 grams) of placebo mixed in 10-12 ounces of a cold beverage to taste preference consumed orally twice daily between meals for 1 week before surgery up until 2 weeks after surgery.
  Active ingredients: alanine
  Interventions: Dietary Supplement: Alanine

INTERVENTIONS:
Dietary Supplement: Essential amino acids — Twice daily consumption for two weeks before and one week after surgery.
  Arms: Treatment
Dietary Supplement: Alanine — Twice daily consumption for two weeks before and one week after surgery.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to prospectively evaluate the effects of essential amino acid (EAA) supplementation on the volume and structure of the muscles surrounding the spine (paraspinal musculature). The main questions it aims to answer are:

* Does EAA supplementation preserve paraspinal muscle volume (PMV) and influence changes to spinal alignment following lumbar spine surgery?
* Does preserving paraspinal muscle volume (PMV) improve post-operative functional status?
* Does preserving PMV reduce post-operative complications, pain, and opioid consumption?

Participants will be asked to:

* Consume either EAA supplement or placebo (alanine) twice daily for one week before and two weeks after lumbar spine surgery
* Record pain levels and medication use in a diary
* Perform functional assessments at routine follow-up visits after surgery
* Undergo blood draws to monitor nutrition status and health
* Undergo one spine magnetic resonance imaging (MRI) before surgery as part of routine surgical planning
* Undergo one additional spine MRI after surgery to monitor PMV after treatment

Researchers will compare the group that consumed EAA supplement and the group that consumed placebo to see if there is a difference in paraspinal muscle volume changes and measures of spinal alignment, functional abilities, pain levels, and opioid use.

DETAILED DESCRIPTION:
This study is a randomized, placebo-controlled, double-blinded, single-center clinical trial to elucidate the effects of perioperative essential amino acid nutritional supplementation in pursuit of the following aim and covariates:

Specific Aim 1: Preserve paraspinal muscle volume and assess impact on spine sagittal balance through measurement of radiographic parameters. Paraspinal muscle atrophy following lumbar spine surgery has been correlated with worse clinical outcomes. It is still not understood whether iatrogenic denervation, immobilization, or nutritional deficiencies lead to the reduced volume in the paraspinal muscles. Investigators will utilize pre- and post-operative MRI scans to quantify changes in paraspinal and psoas muscle cross-sectional area and fatty infiltration, and measure sagittal vertical axis, pelvic incidence, lumbar lordosis, and pelvic tilt, as muscle quality has been correlated with spine balance and degeneration, as well as bone quality.

Specific Aim 2: Assess clinical outcomes postoperatively to determine any possible effect of paraspinal muscle volumes on variability in functional status. Functional assessments will be made using established, validated clinical outcomes measures at baseline and up to 2 years postoperatively. Postoperative adverse events will be recorded throughout the duration of the study, as well as markers of nutritional status using a validated dietary questionnaire and blood sampling. Results will be compared between treatment and control groups to determine if functional status is associated with variability in outcomes related to preservation of native paraspinal muscle volume postoperatively.

Specific Aim 3: Evaluate postoperative pain and opioid consumption postoperatively to determine any possible effect of pain on variability in paraspinal muscle volumes. Patient-reported pain and opioid consumption will be evaluated perioperatively with a daily pain diary, clinician-administered pain assessments, and review of the state-controlled substances database (CURES). Pain ratings, mean morphine equivalents, time to baseline preoperative opioid consumption, and time to opioid discontinuation will be compared between treatment and control groups to determine any relationship between postoperative pain levels on variability in outcomes related to preservation of native paraspinal muscle volume following surgery.

Description of Procedures:

Study team members will review the patient medical record for the minimal amount of health information necessary to determine eligibility in the study prior to obtaining informed consent. Patients undergoing lumbar spine surgery that meet eligibility requirements-determined using standard nutritional and lumbar surgical clinical research inclusion/exclusion criteria applied according to the judgment of the investigator-will receive standardized written and verbal information about the trial from the investigators listed in the study team. For non-English speaking participants, an interpreter will be involved in the consenting process.

A member of the research team will be unblinded and responsible for block randomization of participants with 1:1 allocation to EAA and placebo groups (N=44 each group) using Excel 2016 (Microsoft). The University of California Irvine (UCI) Investigational Drug Services Pharmacy (IDS Pharmacy) is responsible for receiving, labeling, storing, and distributing the products and will collect product containers/any unused products at the conclusion of the supplement period as outlined in the study protocol. The remainder of the study team (including the primary investigator and co-researchers) and the statistician responsible for data analysis will be blinded to randomization.

Demographic and baseline information regarding nutritional, functional, and frailty status will be collected at the baseline visit within 6 weeks to 1 week prior to surgery, including ambulatory status (independent, cane, walker, wheelchair); food preferences (omnivorous, pescatarian, vegan, vegetarian); Protein Screener 55+ (a validated questionnaire to screen for low dietary protein intake in the elderly); modified Fragility Index (a validated risk stratification tool in lumbar spine surgery); and baseline labs (including serum albumin, prealbumin, and transferrin as markers of nutritional status and inflammation), functionality, pain scores, and medication use. From 1 week prior to surgery until 2 weeks postoperatively, patients will consume either a commercially available EAA supplement-containing L-leucine (3.6g), L-lysine as L-lysine HCl (3.2g), L-phenylalanine (3.2g), L-valine (2.4g), L-threonine (2.8g), L-isoleucine (2.0g), L-methionine (0.6g), and L-histidine as L-histidine HCl (2.2g) (Joint Replacement; Mend Labs, New York, NY) twice daily-or calorically-equivalent placebo (alanine, 20g twice daily).

Fellowship-trained spine surgeons will perform all lumbar decompression and/or fusion surgeries using the same posterior operative approach and instrumented fusion of unstable segments if clinically indicated. All patients are hospitalized from the day of surgery until discharge, with the total length of stay dependent on postoperative pain control and progress in physical therapy. Patient-reported pain will be evaluated with a daily pain diary using the Numerical Pain Rating Scale beginning 1 week prior to surgery for at least 2 weeks postoperatively or until termination of opioid consumption (for a maximum of 1 month). Patients will be educated to also record pain levels each time they take an opioid. Opioid consumption-including oxycodone, hydrocodone, morphine, codeine, fentanyl, hydromorphone, and tramadol-will be captured simultaneously through a pain medication diary and compared between treatment groups as mean morphine equivalents. Time to less than baseline opioid consumption and time to opioid discontinuation will also be compared between treatment groups. Clinician-administered patient pain ratings using the Visual Analogue Score will be recorded at baseline, on the day of surgery, and at each postoperative visit.

Timeline of Study Procedures:

1. Screening visit within 6 months to 6 weeks prior to surgery date: consent, physical exam, pregnancy test if appropriate, review of lumbar MRI (approximately 1 hour)
2. Preoperative visit within 6 weeks to 1 week prior to surgery: physical exam, baseline labs, baseline functional mobility and pain assessment, CURES database review, patient education on self-reporting pain, opioid consumption, consumption of other medications, and EAA supplementation or placebo consumption (approximately 2 hours). EAA and placebo will be provided by the manufacturer in the same containers with the same scoop size and the same label instructing patients consume one serving twice a day beginning one before their surgery and for 2 weeks after. These instructions and labels will be provided by Mend and they align with previously studied protocols where the supplement has been fond to be safe. Investigators hope in using the product as directed by Mend to reduce risk for participants and decrease confusion as they can follow the package information.
3. Surgery day (all patients are hospitalized from the day of surgery until discharge, with the total length of stay dependent on postoperative pain control and physical therapy progress). Patients will receive this surgery and the associated postoperative inpatient stay as part of standard of care regardless of their involvement in this study. Research related data collection aside from standard of care during their perioperative inpatient stay will be approximately 1 hour. ( approximately 1 hour)
4. Postoperative follow-up at 2 weeks +/- 5 days: physical exam, functional mobility and pain assessment, labs, review of patient-reported daily pain levels, review of CURES and opioid/medication consumption, review of patient-reported EAA supplementation or placebo consumption logs (approximately 1 hour)
5. Postoperative follow-up at 6-8 weeks +/- 5 days: physical exam, functional mobility and pain assessment, labs, review of CURES and opioid/medication consumption (approximately 30 minutes)
6. Postoperative lumbar MRI without contrast obtained at 8-10 weeks (1 hour)
7. Postoperative follow-up at 12 weeks +/- 5 days: physical exam, review MRI results, functional mobility and pain assessment, review of CURES and opioid/medication consumption (approximately 1 hour)

Statistical Plan:

Power analysis: Sample size analysis was performed a priori using data from the literature evaluating muscle atrophy with and without nutritional supplementation in patients with total knee arthroplasty, as there is no data assessing paraspinal muscle volume after lumbar spine surgery, with an expected difference in primary outcome measure of 4.9% (13.4% +/- 1.9% in control and 8.5% in experimental). Using two independent groups, a continuous variable primary endpoint, an assumed 2-tailed type-1 error rate of 0.05, and a power value of 80% we require a minimum total of 88 patients with 44 in each group.

Overall: Baseline characteristics will be compared between the groups using independent t tests (or the Wilcoxon rank sum test, if the characteristics were not normally distributed) for continuous measures and the chi-square test for categorical measures. Continuous variables will be described using the mean and standard deviation. Categorical variables will be described using absolute frequencies. Pearson's correlation coefficient (r) will be used to assess relationships between paraspinal muscle CSA, opioid consumption as morphine milligram equivalents (MME), clinical functional outcome measures, and postoperative complications. A two-way repeated measured analysis of variance (ANOVA) will evaluate chronological changes in continuous variables between the two groups. Significance will be set at p < 0.05.

Specific Aim 1: Axial T2-weighted lumbar spine MRI at the levels of the L1-5 intervertebral discs using a 3 Tesla (3T) MRI with a phased-array surface coil will be completed within 6 months to 6 weeks (about 1 and a half months) prior to surgery and prior to treatment intervention and will be compared to the repeat MRI completed at 8-10 weeks postoperatively. Bilateral paraspinal muscle cross-sectional area (CSA) will be measured by two experienced musculoskeletal radiologists marking the borders of these muscles. Proton density fat fraction will be used to quantify the proportion of fatty infiltration and overall atrophy will be qualitatively rated based on visual assessment using a visual scale modified from the Goutallier grading system. Sagittal spinopelvic alignment parameters including sagittal vertical axis, pelvic incidence, lumbar lordosis, and pelvic tilt will be measured on both the pre and postoperative MRIs. The intraclass correlation coefficient for this measurement will be evaluated and interpreted according to the predetermined guidelines.

Specific Aim 2: Functional status will be assessed for each treatment arm at baseline, 2 weeks, 6 weeks, and 3 months postoperatively using established, validated clinical outcome measures completed with a trained member of research staff: the Oswestry Disability Index 2.1A, 36-Item Short Form Health Survey (SF-36), Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function, EuroQol-5 Dimension 5 Levels (EQ-5D-5L), 6-minute walk test, and 5 repetitive sit to stand test. Preoperative mortality and morbidity risk will be controlled between treatment groups using the modified Frailty Index. Postoperative adverse events will be recorded throughout the duration of the study, including but not limited to hospital length of stay, surgical site infections, unplanned reoperation, mortality, and medical complications requiring intervention.

Specific Aim 3: Patient-reported pain will be evaluated with a daily pain diary using the Numerical Pain Rating Scale beginning 1 week prior to surgery for at least 2 weeks postoperatively or until termination of opioid consumption (for a maximum of 1 month). Patients will be educated to also record pain levels each time they. Opioid consumption-including oxycodone, hydrocodone, morphine, codeine, fentanyl, hydromorphone, and tramadol-will be captured simultaneously through a pain medication diary and compared between treatment groups as MME.

Safety Monitoring:

A Data Safety Monitoring Board (DSMB) consisting of 7 UCI faculty members from various relevant disciplines-including orthopaedic surgery, anesthesiology, nutrition, pharmacology, biostatistics-has been assembled to ensure the safety of all study participants throughout the duration of the study period. At the first safety meeting prior to subject enrollment, the DSMB will discuss the protocol and agree upon guidelines to study monitoring. Subsequently, study data will be evaluated continuously by the study team and meetings of the DSMB will be held at least two times a year (every 6 months). As part of the purpose of the study is to evaluate the impact of amino acid supplementation on functional/clinical outcomes, pain, and opioid use, data ensuring compliance in supplement ingestion, pain levels, medication use, functional outcomes, and adverse events will be continuously documented. No adverse outcomes are expected given that the amino acid supplement is commercially available and has shown to be safe for human consumption. However, unscheduled emergency meetings may be called at any time by the DSMB or the study investigators should participant safety questions or other unanticipated problems or adverse events arise-such as renal failure, severe GI distress, or melena. Safety updates and reports will be submitted to the UCI Institutional Review Board with the continuing application each year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lumbar pathology requiring lumbar spine surgery without previous surgical intervention
* Failure of more conservative treatment options
* If undergoing fusion, surgery consists of short segment fusion of less than or equal to 5 levels without staged surgery
* Provided voluntary written informed consent to participate in the study
* Able to comply with all study procedures, including taking the assigned treatment or placebo as instructed and attending follow-up visits
* No restrictions on the use of nutritional supplements or dietary modifications
* Able to complete self-report questionnaires and assessments as required by the study protocol
* Confirmed ambulatory status prior to surgery

Exclusion Criteria:

* Comorbidities excluding the use of the proposed nutritional supplement or resulting in decreased serum albumin levels (phenylketonuria, galactosemia, nephrotic syndrome)
* Diagnosis other than lumbar spine pathology requiring lumbar spine surgery
* Non-ambulatory status
* Uncontrolled endocrine disease; heart, kidney, liver, blood, or respiratory disease; peripheral vascular disease
* Unable or unwilling to comply with study procedures, including taking the assigned treatment or placebo as instructed and attending follow-up visits.
* History of congenital metabolic disease (e.g Hartnup disease, Phenylketonuria)
* Active cancer
* Active infection
* Prior protein-calorie supplementation for other clinical indications
* Recent treatment with anabolic steroids or oral corticosteroids for >1 week
* History of chronic opioid consumption > 6 months
* Testosterone or Androgen Supplementation
* History of major head trauma
* Pregnant/breastfeeding women
* History of dementia
* Vulnerable populations (minors, prisoners)
* Lack of decision making capacity
* BMI <18 or > 40
* HbA1c > 7.0
* Patients with pacemakers
* Specific dietary restrictions or allergies that prevent the use of nutritional supplements or dietary modifications
* Currently enrolled in another clinical trial involving interventions that may interfere with the outcomes of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Paraspinal muscle volume | Preoperative lumbar MRI at 6 months-6 weeks prior to surgery, postoperative lumbar MRI at 8-10 weeks after surgery.
  Quantification of bilateral paraspinal muscle cross-sectional area in cm^2 measured with Visage Imaging (San Diego, California) software by two experienced musculoskeletal radiologists marking the borders of these muscles at a standardized spinal level in the lumbar spine. Psoas muscle cross-sectional areas and body height will be used for standardization of body type. Intraclass correlation coefficient between observers will be evaluated and interpreted according to the following guidelines: 0-0.40 poor; 0.41-0.60, moderate; 0.61-0.80, good; and 0.81-1.00 excellent.

SECONDARY OUTCOMES:
Percentage of paraspinal muscle fatty infiltration | Preoperative lumbar MRI at 6 months-6 weeks prior to surgery, postoperative lumbar MRI at 8-10 weeks after surgery.
  Quantification of the proportion of fat to total paraspinal muscle cross-sectional area on MRI proton density fat fraction in ImageJ (National Institutes of Health) by two experienced musculoskeletal radiologists marking the borders of these muscles at a standardized spinal level in the lumbar spine. Intraclass correlation coefficient between observers will be evaluated and interpreted according to the following guidelines: 0-0.40 poor; 0.41-0.60, moderate; 0.61-0.80, good; and 0.81-1.00 excellent.
Paraspinal muscle qualitative fatty infiltration grading (simplified 3-tier classification) | Preoperative lumbar MRI at 6 months-6 weeks prior to surgery, postoperative lumbar MRI at 8-10 weeks after surgery.
  Qualitative rating of paraspinal muscle fatty infiltration by two experienced musculoskeletal radiologists using MRI proton density fat fraction on Visage Imaging (San Diego, California) software. Visual scale modified from the Goutallier grading system: 0 = <10% fat, 1 = <50% fat, 2 = >50% fat. Intraclass correlation coefficient between observers will be evaluated and interpreted according to the following guidelines: 0-0.40 poor; 0.41-0.60, moderate; 0.61-0.80, good; and 0.81-1.00 excellent.
Sagittal spinopelvic alignment (angles measured in degrees) | Preoperative lumbar MRI at 6 months-6 weeks prior to surgery, postoperative lumbar MRI at 8-10 weeks after surgery.
  Radiographic measurements of sagittal vertical axis, pelvic incidence, lumbar lordosis, and pelvic tilt on Visage Imaging (San Diego, California) software. Intraclass correlation coefficient between observers will be evaluated and interpreted according to the following guidelines: 0-0.40 poor; 0.41-0.60, moderate; 0.61-0.80, good; and 0.81-1.00 excellent.
Low back pain (Oswestry disability index 2.1A, total score) | Baseline visit (6 weeks-1 week preoperatively) and 2-week, 6-week, and 12-week follow up visits.
  Validated, 10-item questionnaire for self-reported low back pain and limitations when performing daily activities.
Health-related quality of life (36-Item Short Form Health Survey total and subsection scores) | Baseline visit (6 weeks-1 week preoperatively) and 2-week, 6-week, and 12-week follow up visits.
  Validated, 36-item questionnaire for self-reported quality of life across 8 subsection domains: general health, physical functioning, role physical, role emotional, social functioning, mental health, bodily pain, and vitality.
Self-reported capability to perform activities (PROMIS Physical Function total score) | Baseline visit (6 weeks-1 week preoperatively) and 2-week, 6-week, and 12-week follow up visits.
  Validated questionnaire assessing physical capability to perform activities of daily living and other more strenuous tasks.
Self-reported perceived problems (EuroQol-5 Dimension 5 Levels (EQ-5D-5L) total and subsection scores) | Baseline visit (6 weeks-1 week preoperatively) and 2-week, 6-week, and 12-week follow up visits.
  Validated questionnaire assessing self-reported perceived problems across 5 health state dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression.
6-minute walk test (distance in meters) | Baseline visit (6 weeks-1 week preoperatively) and 2-week, 6-week, and 12-week follow up visits.
  Assessment of cardiopulmonary function and aerobic endurance measured as the distance covered over a 6-minute time frame.
5 repetitive sit-to-stand (time in seconds) | Baseline visit (6 weeks-1 week preoperatively) and 2-week, 6-week, and 12-week follow up visits.
  Assessment of lower extremity functional strength, transitional movements, and balance through timed repetitive sit to stand.
Hospital length of stay (time in days) | Day of surgery until date of discharge
  Time from hospital admission for surgical intervention to discharge.
Incidence of postoperative complications (number of occurrences) | Baseline visit (6 weeks-1 week preoperatively), immediately preoperative on day of surgery, and 2-week, 6-week, and 12-week follow up visits.
  Occurrence of postoperative complications including: surgical site infection, unplanned reoperation, mortality, cardiovascular events, thromboembolism, pneumonia, urinary tract infection, etc.
Self-reported pain levels (Numeric Pain Rating Scale) | Daily recordings starting 1 week prior to surgery up until 2 weeks after surgery or until time of opioid medication discontinuation for a maximum of 1 month after surgery, whichever is sooner.
  Self-recorded pain levels at the time of supplement consumption and at the time of pain medication consumption in a pain diary.
Clinician-administered pain rating (Visual Analog Scale pain score) | Baseline visit (6 weeks-1 week preoperatively), immediately preoperative on day of surgery, and 2-week, 6-week, and 12-week follow up visits.
  Clinician-administered patient pain rating.
Patient-reported pain medication use (measured in mean morphine equivalents) | Starting 1 week prior to surgery up until 2 weeks after surgery or until time of opioid medication discontinuation for a maximum of 1 month after surgery, whichever is sooner.
  Self-recorded pain medication consumption in a pain diary.
Prescription opioid consumption (measured in mean morphine equivalents) | Baseline visit (6 weeks-1 week preoperatively), immediately preoperative on day of surgery, and 2-week, 6-week, and 12-week follow up visits.
  Opioid medication dispensation through clinician monitoring of state controlled substances database (CURES).
Time to opioid discontinuation (time in days) | Day of surgery up until 2 weeks after surgery or until time of opioid medication discontinuation for a maximum of 1 month after surgery, whichever is sooner.
  Time from date of surgery to last use of opioids listed in the self-reported pain diary.
Time to less than baseline opioid consumption (time in days) | Baseline visit (6 weeks-1 week preoperatively) up until 2 weeks after surgery or until time of opioid medication discontinuation for a maximum of 1 month after surgery, whichever is sooner.
  Time to postoperative opioid consumption in mean morphine equivalents less than that measured at baseline (6 weeks to 1 week preoperatively) to day before surgery using the self-reported pain diary.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No